CLINICAL TRIAL: NCT05136430
Title: A Multiple Health Behavior Change Intervention for Overweight and Obese Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cara Murphy, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1608001567; K23DA045078 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-11-29 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation; Obesity
Keywords: smoking; smoking cessation; smoking treatment; quitting smoking; obesity; overweight; multiple health behavior change intervention
MeSH Terms: conditions — Smoking Cessation; Obesity; Smoking; Overweight

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two study conditions at the group level after they have completed baseline assessment. The principal investigator, who is not involved in conducting assessments, will use a random number generator to determine assignment. Participants will learn their condition assignment during their first group session. The interventionist will use a detailed intervention manual to ensure standardization of treatment delivery.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know condition assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Regulation strategies + large changes (SR) (Experimental): This arm will receive the Self-Regulation strategies + large changes (SR) intervention followed by smoking cessation treatment
  Interventions: Behavioral: Self-Regulation strategies + large changes (SR); Other: Smoking Cessation Treatment
- Healthy Lifestyle Education (LE) (Active Comparator): This arm will receive the healthy Lifestyle Education (LE) intervention followed by smoking cessation treatment
  Interventions: Behavioral: Healthy Lifestyle Education (LE); Other: Smoking Cessation Treatment

INTERVENTIONS:
Behavioral: Self-Regulation strategies + large changes (SR) — The first 8 weeks (weeks 1-8) of the 16-week program will include weekly group sessions focused on teaching self-regulation and efforts to produce a 10 lb weight loss to buffer against anticipated post-cessation weight gain. Participants will be taught the core self-regulation skills for controlling their weight. In order to produce an initial weight loss buffer, they will be instructed to self-monitor their intake, given a daily calorie goal, and taught strategies for reducing caloric intake. Structured physical activity, such as brisk walking will also be prescribed and self-monitored. During smoking cessation treatment (weeks 9-16), participants will be asked to continue to use self-regulation skills for monitoring their weight and to use a color zone system (red, yellow, green) to determine what course of action to follow based on whether changes in weight have occurred.
  Arms: Self-Regulation strategies + large changes (SR)
Behavioral: Healthy Lifestyle Education (LE) — The first 8 weeks (weeks 1-8) of the 16-week program will include weekly group sessions focused on living a healthy lifestyle. Information provided will include education on why weight gain happens while quitting smoking, principles of healthy eating (e.g., simple versus complex carbohydrates), physical activity guidelines, and other topics related to living a healthy lifestyle. Participants can choose to use the healthy lifestyle information and education provided however they would like. Participants will not be asked to use self-regulation strategies during either part of the 16-week program.
  Arms: Healthy Lifestyle Education (LE)
Other: Smoking Cessation Treatment — The second 8 weeks (weeks 9-16) of the 16-week program will include weekly group counseling sessions focused on smoking cessation. The smoking cessation treatment provided will be the same in both arms of the study. In preparation of quitting, nicotine replacement therapy lozenges will be provided for 3 weeks prior to quitting (weeks 6-8). A group quit day will occur on week 9. During the smoking cessation portion of treatment (weeks 9-16), participants will be provided with combination nicotine replacement therapy (patches + lozenges) and daily supportive text messages.

SUMMARY:
The purpose of this study is to determine the efficacy, acceptability, and feasibility of an intervention that provides a behavioral weight gain prevention intervention in advance of smoking cessation treatment in individuals with overweight or obesity who smoke cigarettes. The primary aim of this study is to determine feasibility and acceptability and initial efficacy regarding whether preceding 8 weeks of smoking cessation treatment with 8 weeks of self-regulation strategies + large changes for weight gain prevention (SR), compared to 8 weeks of healthy lifestyle education (LE), will result in greater smoking cessation and reduced weight gain. Secondary aims are to study effects on self-efficacy for managing weight and for quitting smoking, negative affect, and delayed reward discounting. Methods: Individuals with overweight or obesity who smoke cigarettes will participate in a 16-week group-based multiple health behavior change intervention. Groups will be randomly assigned to receive either 8 weeks of SR followed by 8 weeks of smoking cessation treatment or 8 weeks of LE followed by 8 weeks of smoking cessation treatment. Smoking cessation treatment in both conditions will include counseling and combination nicotine replacement therapy (patch + lozenges), with a quit day at week 9 of the 16-week intervention. Assessments will occur at baseline, on quit day and 1, 2, and 3 months later. Determining the viability of this strategy in terms of effects on both smoking and weight has high significance to public health.

DETAILED DESCRIPTION:
Aims - The specific aims are to examine: (1) the feasibility, acceptability, and initial efficacy of using self-regulation strategies for weight gain prevention (SR), relative to the provision of healthy lifestyle education (LE), prior to smoking cessation treatment in a pilot study; (2) compare the effect of self-regulation strategies for weight gain prevention (SR), relative to the provision of healthy lifestyle education (LE), prior to smoking cessation treatment, on mechanisms thought to underlie smoking abstinence. Mechanisms include self-efficacy for managing weight and for quitting smoking, negative affect, and delayed reward discounting.

Methodology - A randomized trial will be used to test the feasibility, acceptability, and initial efficacy of using self-regulation strategies for weight gain prevention prior to smoking cessation treatment. Eligible participants will complete baseline assessment and be randomly assigned to one of two conditions. Participants assigned to the SR condition will receive 8 weeks of self-regulation strategies + large changes for weight gain prevention, followed by 8 weeks of smoking cessation treatment. Participants assigned to the LE condition will receive 8 weeks of healthy lifestyle education, followed by 8 weeks of smoking cessation treatment. The intervention will be delivered using a group-based format and will last 16 weeks. Random assignment will occur at the group level. Participants will receive nicotine replacement therapy and counseling as part of the smoking cessation intervention and will quit smoking as a group halfway through treatment (week 9). Assessments will occur at baseline, on quit day (week 9), 1 month after quit day (week 13), 2 months after quit day (week 17), and 3 months after quit day (week 21). Approximately 30 participants will be assigned to each condition (study N=60).

Participant Population - Individuals with overweight or obesity who smoke cigarettes

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2
* smoked ≥ 5 cigarettes/day during the past year
* self-reported motivation to quit smoking
* self-reported desire to prevent or minimize weight gain during smoking cessation
* ability to understand informed consent
* access to a smartphone or tablet

Exclusion Criteria:

* current smoking cessation or weight loss treatment/medication
* more than 1 day/week use of tobacco or nicotine from sources other than cigarettes (other than non-daily use of e-cigarettes in addition to combustible cigarettes)
* weight loss of 20 lbs or more within the past 6 months
* self-reported diagnosis or treatment for an alcohol or substance use disorder within the past 6 months (with the exception of maintenance therapies)
* endorsing recent symptomology suggestive of an eating disorder, an alcohol or substance use disorder, severe depression, or suicidal ideation
* self-reported diagnosis or treatment or evidence of an eating disorder or severe psychiatric disorder (e.g., schizophrenia or bipolar disorder)
* not stabilized on psychotropic medications
* current use of medications known to interact with smoking cessation
* clinically significant medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-Regulation Strategies + Large Changes (SR): Self-Regulation strategies + large changes (SR) arm Weeks 1-8 of the 16-week program will include weekly group sessions focused on teaching self-regulation and efforts to produce weight loss to buffer against anticipated post-cessation weight gain. Participants will be taught the core self-regulation skills for controlling their weight. To produce an initial weight loss buffer, they will be instructed to self-monitor their intake, given a daily calorie goal, and taught strategies for reducing caloric intake. Structured physical activity, such as brisk walking, will also be prescribed and self-monitored. During smoking cessation treatment (weeks 9-16), participants will be asked to continue to use self-regulation skills for monitoring their weight and to use a color zone system (red, yellow, green) to determine what course of action to follow based on whether weight changes have occurred.
  Smoking Cessation Treatment: Weeks 9-16 of the 16-week program will include weekly group counseling sessions focused on smoking cessation. The smoking cessation treatment provided will be the same in both study arms. In preparation of quitting, nicotine replacement lozenges will be provided for 3 weeks prior to quitting (weeks 6-8). A group quit day will occur on week 9. During the smoking cessation portion of treatment (weeks 9-16), participants will be provided with combination nicotine replacement therapy (patches + lozenges) and daily supportive text messages.
Period: Overall Study
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Started | 27 | 28
Completed | 25 | 27
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE) | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 48
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (10.7) | 51.3 (11.7) | 50.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 8 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 12 | 17
  White | 20 | 16 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — region of enrollment (country)
  Participants
    United States | 27 | 28 | 55
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] | 14.6 (5.8) | 14.1 (6.7) | 14.4 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 7-day Point-prevalence Abstinence From Smoking
Description: The number of participants with biochemically-verified 7-day-point prevalence abstinence from smoking
Time Frame: 2 months post-quit (end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 25 | 27
Participants | 11 | 13

2. Primary Outcome: Weight Change
Description: body weight (lbs)
Time Frame: change in weight from baseline to 2 months post-quit (end of treatment)
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 25 | 27
pounds | -5.3 (9.4) | .03 (9.8)

3. Primary Outcome: Treatment Attendance
Description: The percentage of treatment sessions attended through week 10 (one week post-quit) will be used as a measure of attendance to demonstrate feasibility and acceptability
Time Frame: Treatment weeks 1-10
Measure: Mean (Standard Deviation); unit: percentage of sessions
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 27 | 28
percentage of sessions | 85.2 (26.1) | 90.7 (17.2)

4. Secondary Outcome: Number of Participants With 7-day Point-prevalence Abstinence From Smoking
Description: Number of participants with biochemically-verified 7-day-point prevalence abstinence from smoking
Time Frame: 1 months post-quit (end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 26 | 27
Participants | 13 | 13

5. Secondary Outcome: Number of Cigarettes Smoked/Day
Description: Timeline Follow Back (TLFB) interview will assess self-reported number of cigarettes smoked each day, summed over past 28 days
Time Frame: 2 months post-quit (end of treatment)
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 25 | 27
cigarettes per day | 1.9 (3.4) | 1.6 (3.2)

6. Secondary Outcome: Number of Participants Achieving ≥50% Reduction in Cigarettes Per Day Smoked
Description: The number of participants for whom the number of cigarettes smoked per day in the past 7 days has decreased by ≥50%, relative to the number of cigarettes the participant smoked per day at baseline.
Time Frame: 2 months post-quit (end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 25 | 27
Participants | 24 | 26

7. Secondary Outcome: Duration of Longest Period of Abstinence From Smoking
Description: Timeline Follow Back (TLFB) interview will assess self-reported smoking abstinence each day. The longest number of contiguous abstinence days will be recorded starting at quit day.
Time Frame: 2 months post-quit (end of treatment)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 25 | 27
days | 29.1 (22.0) | 40.5 (17.5)

8. Other Pre Specified Outcome: Self-efficacy for Quitting Smoking
Description: The Smoking Self-Efficacy Questionnaire will be used to compare baseline to quit day. Scores range from 12 to 60; higher scores indicate a better outcome.
Time Frame: week 9 (quit day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 26 | 27
score on a scale | 45.0 (10.9) | 45.7 (8.3)

9. Other Pre Specified Outcome: Study Retention
Description: The percentage of participants completing the final outcome assessment will be used to determine study retention.
Time Frame: 3 months post-quit (end of study)
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 27 | 28
Participants | 25 | 27

10. Other Pre Specified Outcome: Self-efficacy for Weight Management After Quitting Smoking
Description: The Weight-Efficacy After Quitting scale will be used to compare baseline to quit day. Scores range from 6 to 60; higher scores indicate a better outcome.
Time Frame: week 9 (quit day)
Measure: Mean (Standard Deviation); unit: score on a scale of self-efficacy
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 26 | 27
score on a scale of self-efficacy | 7.1 (1.4) | 6.4 (1.7)

11. Other Pre Specified Outcome: Delay Discounting
Description: The Monetary Choice Questionnaire will be used to determine a person's rate of impulsive choices when asked to choose between hypothetical amounts of money. Participants will choose between (hypothetical) smaller amounts of money available today or larger amounts of money available following a delay. Responses on this questionnaire are used to determine a person's discount rate, symbolized by the parameter "k", which refers to how steeply delay reduces the value of a reward. Higher k values indicate greater impulsivity (i.e., a greater preference for smaller rewards available immediately than larger rewards available after a delay).
Time Frame: week 9 (quit day)
Measure: Mean (Standard Deviation); unit: k value
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 26 | 26
k value | .037 (.06) | .032 (.07)

12. Other Pre Specified Outcome: Negative Affect Score
Description: Negative affect (i.e., negative emotional states) will be assessed using a measure called the Positive and Negative Affective Schedule (PANAS). This measure is used to derive a "Negative Affect Score." This score is the sum of all items assessing negative affect. The Negative Affect Score can range from 10-50. Higher scores represent more negative affect.
Time Frame: week 9 (quit day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 26 | 27
score on a scale | 17.4 (8.9) | 19.3 (8.0)

13. Other Pre Specified Outcome: Treatment Satisfaction
Description: Treatment satisfaction during the first half of treatment will be assessed via a questionnaire, with higher scores (1-5) indicating greater satisfaction.
Time Frame: week 9 (quit day)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
Number analyzed (Participants) | 26 | 27
score on a scale | 4.5 (.91) | 4.7 (.54)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, approximately 21 weeks
Arm/Group | Self-Regulation Strategies + Large Changes (SR) | Healthy Lifestyle Education (LE)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT05136430/Prot_SAP_000.pdf